CLINICAL TRIAL: NCT04527380
Title: Multicenter, Open-label, Efficacy, Safety, Tolerability, and Pharmacokinetic Study of Subcutaneous Ixekizumab With Adalimumab Reference Arm, in Children With Juvenile Idiopathic Arthritis Subtypes of Enthesitis-related Arthritis (Including Juvenile-Onset Ankylosing Spondylitis) and Juvenile Psoriatic Arthritis
Brief Title: A Study of Ixekizumab (LY2439821) in Children With Juvenile Idiopathic Arthritis Categories of Enthesitis-related Arthritis (Including Juvenile Onset Ankylosing Spondylitis) and Juvenile Psoriatic Arthritis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16694; I1F-MC-RHCG (Other: Eli Lilly and Company); 2018-000681-10 (EudraCT Number); 2023-507184-19-00 (EU CTIS Number)
Record Dates: First submitted 2020-08-24; First posted 2020-08-26 (Actual); Results first posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Juvenile Psoriatic Arthritis; Enthesitis Related Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — ixekizumab; Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ixekizumab - OLT Period (Experimental): Participants received subcutaneous (SC) ixekizumab from week 0 to week 16, following dosing regimens based on body weight:
  * Greater than (>) 50.0 kg: Starting dose 160 mg at week 0, then 80 mg SC every 4 weeks (Q4W) from week 2 to week 16.
  * 25.0-50.0 kg: Starting dose 80 mg at week 0, then 40 mg SC Q4W from week 2 to week 16.
  * 10.0 to less than (<) 25.0 kg: Starting dose 40 mg at week 0, then 20 mg SC Q4W from week 2 to week 16.
  Interventions: Drug: Ixekizumab
- Adalimumab - OLT Period (Active Comparator): Participants received SC adalimumab from week 0 to week 16, following dosing regimens based on body weight:
  * Greater than or equal to (≥) 30.0 kg: 40 mg SC every 2 weeks (Q2W).
  * 10.0 to <30.0 kg: 20 mg SC Q2W.
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Ixekizumab — Administered SC
  Other Names: LY2439821
  Arms: Ixekizumab - OLT Period
Drug: Adalimumab — Administered SC
  Arms: Adalimumab - OLT Period

SUMMARY:
The reason for this study is to see if the study drug ixekizumab is safe and effective in children with juvenile idiopathic arthritis (JIA) categories of enthesitis-related arthritis (ERA) (including juvenile onset ankylosing spondylitis [JoAS]) and juvenile psoriatic arthritis (JPsA).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have active juvenile idiopathic arthritis (categories of enthesitis related arthritis or juvenile psoriatic arthritis)
* Participants must have weight of at least 10 kilograms (Kg), age starting at 2 years for participants with juvenile psoriatic arthritis and starting at 6 years for participants with enthesitis related arthritis
* Participants must have all immunizations up-to-date in agreement with current immunization guidelines, in the opinion of the investigator

Exclusion Criteria:

* Participants must not have active or history of inflammatory bowel disease
* Participants must not have active uveitis
* Participants must not have active or latent tuberculosis
* Participants must not have an active infection
* Participants must not have concurrent use of biologic agents for the treatment of the juvenile idiopathic arthritis

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2028-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM -5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (43):
- Argentina (2):
  - Instituto CAICI SRL Loc. 15, Rosario, Santa Fe Province
  - Centro Medico Privado de Reumatologia Loc. 20, San Miguel de Tucumán, Tucumán Province
- Belgium (3):
  - Cliniques universitaires Saint-Luc, Brussels, Bruxelles-Capitale, Région de
  - UZ Gent, Ghent, Oost-Vlaanderen
  - UZ Leuven, Leuven, Vlaams-Brabant
- Czechia (3):
  - Oddeleni revmatologie deti a dospelych Loc. 1, Prague, Praha 5
  - Dětská klinika Loc. 11, Olomouc
  - Klinika detskeho a dorostoveho lekarstvi Loc. 1, Prague
- Aarhus Universitetshospital, Skejby, Aarhus, Central Jutland, Denmark
- France (5):
  - Service rhumatologie Loc., Bron, Auvergne-Rhône-Alpes
  - Service de consultation pédiatrique Loc. 1, Montpellier, Hérault
  - Rhumatologie pediatrique et CEREMAIA Loc. 1, Le Kremlin-Bicêtre, Paris
  - RHUMATOLOGIE Loc. 1, Poitiers, Vienne
  - Centre d'Investigation Clinique Loc. 1, Paris
- Germany (7):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Asklepios Klinik Sankt Augustin, Sankt Augustin, North Rhine-Westphalia
  - St. Josef-Stift Sendenhorst, Sendenhorst, North Rhine-Westphalia
  - Helios Klinikum Berlin-Buch, Berlin
  - Charité Campus Virchow-Klinikum, Berlin
  - Klinikum Bremen-Mitte, Bremen
  - Praxis Kinder- und Jugendrheumatologie Dr. Ivan Foeldvari, Hamburg
- Italy (6):
  - University of Naples Federico II, Napoli, Campania
  - IRCCS Istituto Giannina Gaslini, Genoa, Liguria
  - Centro Specialistico Ortopedico Traumatologico Gaetano Pini - CTO, Milan, Lombardy
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - A.O.Universitaria Meyer, Florence, Tuscany
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
- CITER Centro de Investigación y Tratamiento de las Enfermedades Reumáticas, Mexico City, Mexico City, Mexico
- UMC Utrecht - Wilhelmina Kinderziekenhuis, Utrecht, Netherlands
- Spain (5):
  - Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona [Barcelona]
  - Hospital Infantil Universitario Niño Jesús, Madrid, Madrid, Comunidad de
  - H.R.U Málaga - Hospital Materno-infantil, Málaga
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Switzerland (2):
  - Universitäts-Kinderspital beider Basel, Basel, Canton of Basel-City
  - Ostschweizer Kinderspital, Sankt Gallen
- United Kingdom (7):
  - Bristol Royal Hospital for Children, Bristol, Bristol, City of
  - Alder Hey Children's Hospital, Liverpool, England
  - Queen's Medical Centre, Nottingham University Hospitals, Nottingham, Nottinghamshire
  - Oxford University Hospitals - Nuffield Orthopaedic Centre, Oxford, Oxfordshire
  - Royal Stoke University Hospital, Stoke-on-Trent, Staffordshire
  - Haywood Community Hospital, Stoke-on-Trent, Staffordshire
  - Sheffield Children's Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Ixekizumab (LY2439821) in Children With Juvenile Idiopathic Arthritis Categories of Enthesitis-related Arthritis (Including Juvenile Onset Ankylosing Spondylitis) and Juvenile Psoriatic Arthritis — https://trials.lilly.com/en-US/trial/282976

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The results reported are for the primary outcome up to Week 16 (OLT period); data beyond Week 16 will be reported after study completion, at the time of final results reporting.
Pre-assignment Details: The study was designed to be conducted in four periods: Open Label Treatment (OLT) Period (Week 0-16), Open Label Extension (OLE) Period (Week 16-104), Long Term Extension (LTE) Period (Week 104-264), and a 12-week Post Treatment Follow-Up (PTFU) Period.
Period: Overall Study
Arm/Group | Ixekizumab - OLT Period | Adalimumab - OLT Period
Started (As pre-specified in the statistical analysis plan, all randomized participants were reported, per treatment regimen, as exposure was the same across the different treatment groups.) | 81 | 20
Received at Least One Dose of Study Drug | 81 | 20
Completed | 80 | 19
Not Completed | 1 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: As pre-specified in the statistical analysis plan, all randomized participants were reported, per treatment regimen, as exposure was the same across the different treatment groups.
Groups:
- Ixekizumab - OLT Period: Participants received SC ixekizumab from week 0 to week 16, following dosing regimens based on body weight:
  * > 50.0 kg: Starting dose 160 mg at week 0, then 80 mg SC Q4W from week 2 to week 16.
  * 25.0-50.0 kg: Starting dose 80 mg at week 0, then 40 mg SC Q4W from week 2 to week 16.
  * 10.0 to < 25.0 kg: Starting dose 40 mg at week 0, then 20 mg SC Q4W from week 2 to week 16.
- Adalimumab - OLT Period: Participants received SC adalimumab from week 0 to week 16, following dosing regimens based on body weight:
  * ≥ 30.0 kg: 40 mg SC Q2W.
  * 10.0 to <30.0 kg: 20 mg SC Q2W.
- Total: Total of all reporting groups
Arm/Group | Ixekizumab - OLT Period | Adalimumab - OLT Period | Total
Number analyzed (Participants) | 81 | 20 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.10 (3.07) | 13.30 (3.16) | 13.10 (3.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 8 | 44
  Male | 45 | 12 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 4 | 30
  Not Hispanic or Latino | 26 | 5 | 31
  Unknown or Not Reported | 29 | 11 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 4 | 15
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 69 | 15 | 84
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 8 | 1 | 9
  Belgium | 2 | 1 | 3
  Czechia | 3 | 0 | 3
  France | 3 | 0 | 3
  Germany | 21 | 10 | 31
  Italy | 7 | 0 | 7
  Mexico | 17 | 4 | 21
  Netherlands | 1 | 0 | 1
  Spain | 5 | 0 | 5
  Switzerland | 1 | 1 | 2
  United Kingdom | 13 | 3 | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) 30 (Ixekizumab - OLT Period)
Description: JIA ACR, is comprised of 6 variables: number of active joints, number of joints with limited range of motion, Physician's Global Assessment of Disease Activity, Parent's Global Assessment of Well-Being, physical function (measured by the Childhood Health Assessment Questionnaire [CHAQ]), and acute-phase reactants (high-sensitivity C-reactive protein [hsCRP] and erythrocyte sedimentation rate [ESR]). A JIA ACR30 response is defined as at least 30% improvement from baseline in at least 3 of any 6 variables in the core set, with no more than 1 of the remaining variables worsening by more than 30%.
Time Frame: Week 16
Population: All randomized participants who received at least one dose of study drug. Non responder Imputation (NRI) is applied for inadequate responders and participants who had missing data at Week 16 for any reason including discontinuation. As per the pre-specified statistical analysis plan, outcomes were analyzed and reported by treatment regimen, as exposure was the same across the different treatment groups.
Measure: Number; unit: Percentage of participants
Groups:
- Ixekizumab - OLT Period: Participants received SC ixekizumab from week 0 to week 16, following dosing regimens based on body weight:
  * > 50.0 kg: Starting dose 160 mg at week 0, then 80 mg SC Q4W from week 2 to week 16.
  * 25.0-50.0 kg: Starting dose 80 mg at week 0, then 40 mg SC Q4W from week 2 to week 16.
  * 10.0 to< 25.0 kg: Starting dose 40 mg at week 0, then 20 mg SC Q4W from week 2 to week 16.
Arm/Group | Ixekizumab - OLT Period
Number analyzed (Participants) | 81
Percentage of participants | 88.9

2. Secondary Outcome: Percentage of Participants Achieving JIA ACR 30 (Adalimumab - OLT Period)
Description: as for outcome 1
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Adalimumab - OLT Period
Number analyzed (Participants) | 20
Percentage of participants | 95.0

3. Secondary Outcome: Percentage of Participants Achieving JIA ACR 50/70/90/100 (OLT Period)
Description: JIA ACR, is comprised of 6 core set variables: number of active joints, number of joints with limited range of motion, Physician's Global Assessment of Disease Activity, Parent's Global Assessment of Well-Being, physical function (measured by the Childhood Health Assessment Questionnaire [CHAQ]), and acute-phase reactants (high-sensitivity C-reactive protein [hsCRP] and erythrocyte sedimentation rate [ESR]). A JIA ACR 50/70/90 response is defined as a greater than or equal to (≥) 50/70/90/100% improvement from baseline in at least 3 of any 6 variables in the core set, with no more than 1 of the remaining variables worsening by more than 30%.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Groups:
- Ixekizumab - OLT Period: Participants received SC ixekizumab from week 0 to week 16, following dosing regimens based on body weight:
  -> 50.0 kg: Starting dose 160 mg at week 0, then 80 mg SC Q4W from week 2 to week 16.
  * 25.0-50.0 kg: Starting dose 80 mg at week 0, then 40 mg SC Q4W from week 2 to week 16.
  * 10.0 to < 25.0 kg: Starting dose 40 mg at week 0, then 20 mg SC Q4W from week 2 to week 16.
Arm/Group | Ixekizumab - OLT Period | Adalimumab - OLT Period
Number analyzed (Participants) | 81 | 20
Percentage of participants
  ACR50 response | 79 | 90.0
  ACR70 response | 64.2 | 65.0
  ACR90 response | 29.6 | 40.0
  ACR100 response | 18.5 | 35.0

4. Secondary Outcome: Percentage of Participants Achieving JIA ACR 30/50/70/90/100 (OLE Period)
Description: JIA ACR, is comprised of 6 core set variables: number of active joints, number of joints with limited range of motion, Physician's Global Assessment of Disease Activity, Parent's Global Assessment of Well-Being, physical function (measured by the Childhood Health Assessment Questionnaire [CHAQ]), and acute-phase reactants (high-sensitivity C-reactive protein [hsCRP] and erythrocyte sedimentation rate [ESR]). A JIA ACR 30/50/70/90 response is defined as a greater than or equal to (≥) 30/50/70/90/100% improvement from baseline in at least 3 of any 6 variables in the core set, with no more than 1 of the remaining variables worsening by more than 30%.
Time Frame: Week 104
Reporting Status: Not Posted, anticipated posting 2029-04

5. Secondary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) for Juvenile Psoriatic Arthritis (JPsA) Participants With at Least 3% Body Surface Area (BSA) at Baseline (OLT Period)
Description: The PASI is an index that combines assessments of the extent of body-surface involvement in 4 anatomical regions (head, trunk, arms, and legs) and the severity of scaling (S), redness (R), and plaque induration/infiltration thickness (T) in each region, yielding an overall score of 0 for no psoriasis to 72 for the most severe disease. Severity is rated for each index (R, S, T) on a 0 to 4 scale (0 for no involvement up to 4 for severe involvement):
  0 = none
  1. = slight
  2. = moderate
  3. = severe
  4. = very severe The various body regions are weighted to reflect their respective proportion of BSA.
Time Frame: Baseline, Week 16
Population: All randomized participants who received at least one dose of study drug with baseline psoriatic lesion(s) involving ≥3% BSA. For missing post-baseline values for subjects who discontinued the study drug due to adverse events, imputation was performed using the Modified Baseline Observation Carried Forward (mBOCF) method. As per the pre-specified statistical analysis plan, outcomes were analyzed and reported by treatment regimen, as exposure was the same across the different treatment groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ixekizumab - OLT Period | Adalimumab - OLT Period
Number analyzed (Participants) | 14 | 1
score on a scale | -3.80 (3.541) | -0.70 (NA) — Standard deviation in the adalimumab arm was not estimable due to insufficient data (as only one participant was available for analysis).

6. Secondary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) for Juvenile Psoriatic Arthritis (JPsA) Participants With at Least 3% Body Surface Area (BSA) at Baseline (OLE Period)
Description: as for outcome 5
Time Frame: Baseline, Week 104
Reporting Status: Not Posted, anticipated posting 2029-04

7. Secondary Outcome: Change From Baseline in Leeds Enthesitis Index (LEI) for Participants With Enthesitis Related Arthritis (ERA) at Baseline (OLT Period)
Description: The LEI was developed specifically for use in psoriatic arthritis (PsA). It measures enthesitis at 6 sites (lateral epicondyle of humerus, right/left (R/L); medial femoral condyle, (R/L); Achilles tendon insertion, (R/L)). Each site is assigned a score of 0 (absent) or 1 (present); the results from each site are then added to produce a total score (range 0 to 6) with the higher scores indicating more severe enthesitis.
Time Frame: Baseline, Week 16
Population: All randomized participants who received at least one dose of study drug and had a baseline enthesitis (LEI >0). For missing post-baseline values for subjects who discontinued the study drug due to adverse events, imputation was performed using the Modified Baseline Observation Carried Forward (mBOCF) method. As per the pre-specified statistical analysis plan, outcomes were analyzed and reported by treatment regimen, as exposure was the same across the different treatment groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ixekizumab - OLT Period | Adalimumab - OLT Period
Number analyzed (Participants) | 40 | 4
score on a scale | -1.63 (1.005) | -1.50 (0.577)

8. Secondary Outcome: Change From Baseline in Leeds Enthesitis Index (LEI) for Participants With Enthesitis Related Arthritis (ERA) at Baseline (OLE Period)
Description: as for outcome 7
Time Frame: Baseline, Week 104
Reporting Status: Not Posted, anticipated posting 2029-04

9. Secondary Outcome: Percentage of Participants With Disease Flare (OLT Period)
Description: Disease flare is defined as worsening of ≥30% from baseline in at least 3 of the 6 JIA ACR core set criteria and an improvement of ≥30% in no more than one of the criteria. The JIA ACR, is comprised of 6 core set variables: number of active joints, number of joints with limited range of motion, Physician's Global Assessment of Disease Activity, Parent's Global Assessment of Well-Being, physical function (measured by the Childhood Health Assessment Questionnaire [CHAQ]), and acute-phase reactants (high-sensitivity C-reactive protein [hsCRP] and erythrocyte sedimentation rate [ESR]).
Time Frame: Week 2 through Week 16
Population: All randomized participants, even if the participant does not take the assigned treatment. As per the pre-specified statistical analysis plan, outcomes were analyzed and reported by treatment regimen, as exposure was the same across the different treatment groups.
Measure: Number; unit: Percentage of participants
Arm/Group | Ixekizumab - OLT Period | Adalimumab - OLT Period
Number analyzed (Participants) | 81 | 20
Percentage of participants | 0 | 0

10. Secondary Outcome: Percentage of Participants With Disease Flare (OLE Period)
Description: as for outcome 9
Time Frame: Baseline through Week 104
Reporting Status: Not Posted, anticipated posting 2029-04

11. Secondary Outcome: Pharmacokinetics (PK): Trough Concentrations (C-trough) of Ixekizumab (Ixekizumab - OLT Period)
Description: C-trough were measured at specified time points to assess the minimum concentration of ixekizumab in the blood before the next dose was administered.
Time Frame: Week 4, 12 and 16 : Pre-dose
Population: All randomized participants who received at least one dose of the study drug and had evaluable C-trough data at the specified time points. As per the pre-specified statistical analysis plan, the PK outcome was analyzed and reported for the ixekizumab treatment arm, categorized by weight.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (µg/mL)
Groups:
- Ixekizumab - OLT Period (>50 kg Group): Participants weighing >50.0 kg who received a starting dose of 160 mg at week 0, then 80 mg SC Q4W from week 2 to week 16 were included in this arm.
- Ixekizumab - OLT Period (25 to 50 kg Group): Participants weighing 25.0 to 50.0 kg who received a starting dose of 80 mg at week 0, then 40 mg SC Q4W from week 2 to week 16 were included in this arm.
- Ixekizumab - OLT Period (10 to <25 kg Group): Participants weighing 10.0 to <25.0 kg who received a starting dose of 40 mg at week 0, then 20 mg SC Q4W from week 2 to week 16 were included in this arm.
Arm/Group | Ixekizumab - OLT Period (>50 kg Group) | Ixekizumab - OLT Period (25 to 50 kg Group) | Ixekizumab - OLT Period (10 to <25 kg Group)
Number analyzed (Participants) | 55 | 20 | 6
micrograms per milliliter (µg/mL)
  Week 4 | 4.43 (71) | 5.09 (38) | 3.28 (56)
  Week 12 | 3.25 (68) | 3.39 (57) | 2.95 (41)
  Week 16 | 3.47 (55) | 3.32 (37) | 2.80 (46)

12. Secondary Outcome: Pharmacokinetics (PK): Trough Concentrations (C-trough) of Ixekizumab (Ixekizumab - OLE Period)
Description: as for outcome 11
Time Frame: Week 20, 32, 56, 80 and 104 : Pre-dose
Reporting Status: Not Posted, anticipated posting 2029-04

13. Secondary Outcome: Percentage of Participants With Treatment-emergent Positive Anti-ixekizumab Antibodies (Ixekizumab - OLT Period)
Description: Percentage of participants with treatment-emergent positive anti-ixekizumab antibodies was summarized by treatment group. Percentage was calculated based on the number of evaluable participants and was calculated by number of participants with treatment-emergent positive anti-ixekizumab antibodies / number of evaluable participants * 100%.
Time Frame: Baseline through Week 16
Population: All randomized participants who received at least one dose of the study drug and had evaluable data. As per the pre-specified statistical analysis plan, outcomes were analyzed and reported by treatment regimen, as exposure was the same across the different treatment groups.
Measure: Number; unit: Percentage of participants
Arm/Group | Ixekizumab - OLT Period
Number analyzed (Participants) | 80
Percentage of participants | 8.8

14. Secondary Outcome: Percentage of Participants With Treatment-emergent Positive Anti-ixekizumab Antibodies (Ixekizumab - OLE Period)
Description: as for outcome 13
Time Frame: Baseline through Week 104
Reporting Status: Not Posted, anticipated posting 2029-04

ADVERSE EVENTS:
Time Frame: Baseline up to week 16 (until OLT period)
Description: * All randomized participants who received at least 1 dose of the study drug.
  * As per the pre-specified statistical analysis plan, safety data were analyzed and reported by treatment regimen, as exposure was the same across the different treatment groups.
  * Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | Ixekizumab - OLT Period | Adalimumab - OLT Period
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/20
Serious Adverse Events (participants affected / at risk) | 3/81 | 3/20
Other Adverse Events (participants affected / at risk) | 66/81 | 15/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixekizumab - OLT Period (N=81) | Adalimumab - OLT Period (N=20)
Bicytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Ixekizumab - OLT Period (N=81) | Adalimumab - OLT Period (N=20)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Chalazion (Eye disorders) | 1 (1) | 0 (0)
Eye haematoma (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Retinal degeneration (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 1 (2)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 7 (8) | 0 (0)
Application site pain (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (3) | 0 (0)
Illness (General disorders) | 1 (2) | 0 (0)
Influenza like illness (General disorders) | 2 (2) | 0 (0)
Injection site erythema (General disorders) | 2 (4) | 1 (1)
Injection site haematoma (General disorders) | 1 (1) | 0 (0)
Injection site hypersensitivity (General disorders) | 2 (3) | 0 (0)
Injection site pain (General disorders) | 8 (21) | 0 (0)
Injection site rash (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 13 (29) | 1 (1)
Injection site swelling (General disorders) | 2 (3) | 0 (0)
Injection site urticaria (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Puncture site induration (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 6 (7) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Beta haemolytic streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1)
Covid-19 (Infections and infestations) | 7 (7) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Enterobiasis (Infections and infestations) | 1 (1) | 0 (0)
Fungal foot infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 11 (13) | 4 (6)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Pharyngitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0)
Rhinitis (Infections and infestations) | 5 (6) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 0 (0)
Upper respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 3 (3) | 1 (1)
Viral pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foreign body ingestion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injection related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Atypical lymphocytes increased (Investigations) | 1 (1) | 0 (0)
Blood cholesterol decreased (Investigations) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Blood parathyroid hormone increased (Investigations) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 2 (3) | 0 (0)
C-reactive protein increased (Investigations) | 2 (2) | 0 (0)
Cd4/cd8 ratio decreased (Investigations) | 1 (1) | 0 (0)
Eosinophil count increased (Investigations) | 4 (4) | 0 (0)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
Monocyte count decreased (Investigations) | 1 (1) | 1 (1)
Protein urine present (Investigations) | 1 (1) | 0 (0)
Vitamin d decreased (Investigations) | 2 (2) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Amplified musculoskeletal pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (4) | 1 (1)
Headache (Nervous system disorders) | 13 (20) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Initial insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Tearfulness (Psychiatric disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 1/45 (1) | 0/12 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Allergic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 2 (3)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Endodontic procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Vein disorder (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT04527380/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-12): https://cdn.clinicaltrials.gov/large-docs/80/NCT04527380/SAP_001.pdf